CLINICAL TRIAL: NCT03624166
Title: Impact of Sub-anesthetic Dose of Ketamine on Post Spinal Hypotension in Caesarean Delivery :Prospective , Randomized Double- Blinded Study
Brief Title: Impact of Sub-anesthetic Dose of Ketamine on Post Spinal Hypotension in Caesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FAMUS R 38/ 2018
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Ketamine; Anesthetics, General; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Active Comparator): sub- anesthetic dose of ketamine 0.5 mg/kg will be given in 3 ml volume
  Interventions: Drug: Ketamine
- isotonic saline (Placebo Comparator): isotonic saline 3 ml volume will be given
  Interventions: Drug: isotonic saline

INTERVENTIONS:
Drug: Ketamine — patients will receive sub- anesthetic dose of ketamine 0.5 mg/kg in 3 ml of isotonic saline after spinal anesthesia
  Other Names: general anesthetic
  Arms: Ketamine
Drug: isotonic saline — patients will receive 3 ml of isotonic saline after spinal anesthesia
  Arms: isotonic saline

SUMMARY:
The purpose of this study is to evaluate the effect of sub anesthetic dose of ketamine on vasopressor (Ephedrine) requirement to prevent maternal hypotension after spinal anesthesia in caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Physical status American Society of Anesthesiologist(ASA) I or II. Full term pregnancy

Exclusion Criteria:

* ,Pre-eclampsia.
* Chronic hypertension.
* Cardiovascular troubles.
* any contraindications to spinal anesthesia as back infection , coaguolopathy , patient refusal

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
incidence of hypotension | 5 hours
  after spinal anesthesia sub- anesthetic dose of ketamine will be given and blood pressure will be recorded every 2 minutes till delivery , every 5 minutes till end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt